CLINICAL TRIAL: NCT00930774
Title: Evaluation of Approaches to Auditory Rehabilitation for Mild TBI
Brief Title: Approaches to Auditory Rehabilitation for Mild Traumatic Brain Injury
Acronym: mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: C7054-R; 02386 (Other: Portland VA IRB); 11-1808 (Other: Portland VA IRB)
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; rehabilitation; auditory processing disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Auditory Perceptual Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- FM System (Experimental): Provision of FM assistive device
  Interventions: Device: FM system
- Auditory Training (Experimental): Provision of auditory training
  Interventions: Behavioral: Auditory training
- FM System and Auditory Training (Experimental): Provision of FM assistive device and auditory training
  Interventions: Device: FM system; Behavioral: Auditory training
- Standard-of-Care (No Intervention): Standard-of-care informational counseling

INTERVENTIONS:
Device: FM system — Frequency modulation assistive device
  Arms: FM System; FM System and Auditory Training
Behavioral: Auditory training — Participation in computerized auditory training program for eight weeks
  Arms: Auditory Training; FM System and Auditory Training

SUMMARY:
Many soldiers returning from their recent service in Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) were exposed to blasts during combat. About 60% of blast-injured soldiers are diagnosed with traumatic brain injury (TBI), with approximately 18% having a mild TBI (mTBI). mTBI is associated with many symptoms, including memory problems, headaches, difficulty concentrating, increased anxiety, and, especially relevant here, reports of difficulty understanding speech in noisy environments and/or when people speak rapidly. While problems understanding rapid speech or speech in noise are associated with hearing loss, many of the OIF/OEF veterans with these complaints have clinically normal hearing. Although there is no physical damage to their ears, these veterans' hearing problems have a negative impact on their quality-of-life and functioning. Thus it is incumbent upon the VA to examine intervention approaches for veterans with normal/near-normal auditory sensitivity and significant complaints of difficulty hearing. Currently, there is no standard-of-care for these veterans other than providing information about hearing, hearing conservation, and the use of communication strategies. Two forms of rehabilitation likely to be more effective than such an informational-counseling approach are: (1) the use of personal miniaturized Frequency modulation (FM) systems, and (2) the provision of auditory training with Posit Science Brain Fitness Program (BFP). Personal FM systems increase the loudness of the speech signal relative to that of the unwanted noise, while the BFP training improves the ability to listen by taking advantage of the brain's ability to change (i.e., neural plasticity). In this study veterans will randomly be selected to receive one of four treatments: (1) FM use alone, (2) BFP training alone, (3) FM+BFP training combined, and (4) informational-counseling. The effectiveness of the interventions will be compared using self-report of hearing functioning on standard questionnaires. Results will contribute to the development of evidence-based intervention approaches for blast-exposed veterans with reported functional hearing difficulties and normal/near-normal auditory sensitivity.

DETAILED DESCRIPTION:
The long-term goal of this study is to develop evidence-based auditory rehabilitation for veterans who have normal/near-normal peripheral auditory function and significant complaints of difficulty hearing. Many are veterans of the OIF/OEF conflicts who have been exposed to blast - the most common wounding etiology in these conflicts. Approximately 18% of blast-injured veterans are diagnosed with mild traumatic brain injury (mTBI). mTBI can result in post-concussive symptoms such as memory problems, difficulty concentrating, increased anxiety, and functional hearing difficulties in the presence of clinically-normal hearing sensitivity.

Currently there is no standard-of-care auditory rehabilitation for veterans with normal/near-normal auditory sensitivity and complaints of difficulty hearing. At a minimum, the VA recommends provision of information about the auditory system, hearing conservation and use of communication strategies. Two interventions likely to be more efficacious are: (1) use of personal FM (frequency modulation) systems, and/or (2) auditory training. FM systems are effective for managing auditory problems in children with normal/near normal peripheral hearing. FM systems substantially improve the signal-to-noise ratio of speech in noisy and reverberant environments, theoretically making more resources available for higher level processing. Auditory training takes advantage of neural plasticity. The Posit Science Brain Fitness Program (BFP) is an auditory training program for adults that can improve temporal processing and working memory of older adults. Combining use of FM systems with auditory training has been shown to improve speech understanding and to decrease reported hearing abilities among adults with sensorineural hearing loss and functional hearing complaints.

No study has systemically examined the relative efficacy of FM use and/or auditory training for veterans with mTBI and normal/almost normal hearing sensitivity. The effectiveness of these two intervention strategies will be examined in this study through a between-subjects randomized controlled clinical trial comparing the outcomes of: (1) FM use alone, (2) BFP alone, and (3) FM+BFP combined. All groups will also receive informational-counseling, as will (4) a control group. Outcomes will be measured subjectively through self-report of auditory competence.

The results of the study will help to determine whether or not the use of FM systems or auditory training, either alone or combined, are efficacious interventions for blast-exposed veterans with reported functional hearing difficulties and normal/near-normal auditory sensitivity. Results will contribute to the development of evidence-based auditory rehabilitation for these veterans, moving VA closer to fulfilling its goal of providing excellence in patient care, veterans' benefits and customer satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Participants will be OIF/OEF veterans with no exclusions based on age, ethnicity, or gender. To be included in the study participants will:

* Report difficulty understanding speech in difficult listening environments disproportionate to loss in hearing sensitivity, as defined by self-referral to the study
* Have hearing thresholds <= 65 decibels hearing loss (dB HL) at 0.5, 1.0, 2.0, 3.0 & 4.0 kilohertz (kHz)
* Cognitive abilities sufficient to participate in the study, as determined by an age and education-level appropriate score on the Mini Mental State Exam (MMSE; Folstein, Robins, & Helzer, 1983; Crum et al., 1993),
* English as a first language,
* Openness to using a personal FM system for a four-week period and/or to conducting auditory training over an eight-week period, as determined through interview.

Exclusion Criteria:

* Asymmetric pure tone thresholds (left-right difference > 15 dB HL at frequencies of 500 through 4000 Hz),
* Presence of neurological, psychiatric or physical disorders, or co-morbid diseases that would prevent completion of the study as determined by chart review,
* Best corrected vision worse than 20/63 as measured with the Smith-Kettlewell Institute Low Luminance (SKILL) Card

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Saunders, Principal Investigator — VA Medical Center, Portland
Locations (2):
- United States (2):
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Medical Center, Portland, Portland, Oregon

REFERENCES:
- [Derived] Saunders GH, Frederick MT, Arnold M, Silverman S, Chisolm TH, Myers P. Auditory difficulties in blast-exposed Veterans with clinically normal hearing. J Rehabil Res Dev. 2015;52(3):343-60. doi: 10.1682/JRRD.2014.11.0275. PMID 26237266

RESULTS

PARTICIPANT FLOW:
Groups:
- FM System and Auditory Training: Provision of frequency modulation (FM) assistive device and auditory training
  FM system: Frequency modulation assistive device
  Auditory training: Participation in computerized auditory training program for eight weeks
Period: Overall Study
Arm/Group | FM System | Auditory Training | FM System and Auditory Training | Standard-of-Care
Started | 25 | 25 | 24 | 25
Completed | 24 | 16 | 22 | 25
Not Completed | 1 | 9 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 9 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants were male and female blast-exposed Veterans from the Operation Enduring Freedom/Operation Iraqi Freedom conflicts who reported difficulties hearing speech in noise/when spoken quickly/other difficult circumstances but had clinically-normal hearing.
Groups:
- FM System + Auditory Training: Provision of FM assistive device and auditory training
  FM system: Frequency modulation assistive device
  Auditory training: Participation in computerized auditory training program for eight weeks
- Total: Total of all reporting groups
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-Care | Total
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (7.8) | 33.9 (9.2) | 33.9 (7.7) | 33.7 (8.0) | 34.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 0 | 3 | 11
  Male | 20 | 22 | 24 | 22 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 1 | 4 | 11
  White | 19 | 22 | 21 | 21 | 83
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 4 | 10
  Not Hispanic or Latino | 23 | 23 | 20 | 21 | 87
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Pure tone sensitivity [Mean (Standard Deviation); unit: Decibels hearing level] — Assessment of hearing ability at threshold for frequencies between 250 hertz and 8000 hertz
  Decibels hearing level | 12.3 (6.1) | 12.0 (5.3) | 12.9 (5.4) | 12.1 (4.4) | 12.2 (5.1)
Word recognition score [Mean (Standard Deviation); unit: percent correct] — Assessment of ability to repeat back simple words presented at 40 decibels above threshold
  percent correct | 95.5 (5.8) | 95.2 (5.4) | 97.3 (2.8) | 95.6 (3.9) | 95.9 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Competence Score From the Psychosocial Impact of Assistive Devices Scale (PIADS)
Description: Assesses the impact a rehabilitative intervention has on perceived Competence (perceived functional capability, independence and performance). Responses are reported on a 7-point scale that ranges from -3 (maximum negative impact) to +3 (maximum positive impact). The mid-point, zero, indicates no impact or no perceived change
Time Frame: Immediately post-intervention between weeks 8 and 12
Population: The number of participants analyzed differs from the number of baseline enrollees due to participant attrition. Specifically, one individual in arm 1 (FM system), eleven participants in arm 2 (Auditory training), four in arm 3 (FM system and auditory training) and three in arm 4 (standard of care) chose not to attend the follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
units on a scale | 0.56 (0.55) | .37 (.52) | .62 (.61) | .41 (.76)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.527, ANOVA; df = 3,83; F=0.748

2. Primary Outcome: Stroop Color and Word Test
Description: Measure of processing interference that assesses the ability to cope with cognitive stress and process complex input. It consists of a Word Page with color words printed in black ink, a Color Page with 'Xs' printed in color, and a Color-Word Page with words from the first page printed in colors from the second page (the color and the word do not match). The test-taker looks at each sheet and moves down the columns, reading words or naming the ink colors as quickly as possible within a time limit. Interference raw scores were converted into t-scores for analysis. T-score benefit was the analytic metric used. T-score benefit = post-intervention score minus baseline score
Time Frame: Baseline and Immediately post-intervention (between weeks 8 and 12).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score benefit
Groups:
- FM Sytem + Auditory Training: Provision of FM assistive device and auditory training
  FM system: Frequency modulation assistive device
  Auditory training: Participation in computerized auditory training program for eight weeks
Arm/Group | FM System | Auditory Training | FM Sytem + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
t-score benefit | 1.2 (11.5) | 0.4 (3.0) | 1.1 (5.1) | 1.6 (10.6)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM Sytem + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.835, ANOVA; df = 3,83; F=0.286

3. Secondary Outcome: Hearing in Noise Test
Description: Hearing In Noise Test assesses speech understanding in noise assessed. Sentences are presented in a background of noise. The signal to noise ratio is varied adaptively to obtained the signal to noise ratio at which participants can correctly repeat back 50% of sentences presented in speech-shaped noise is determined. A lower signal to noise ratio indicates better performance.
Time Frame: Immediately post-intervention between weeks 8 and 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Decibels (signal to noise ratio)
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
Decibels (signal to noise ratio) | -8.1 (3.2) | -8.1 (2.0) | -8.2 (4.3) | -7.9 (2.6)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.983, ANOVA; df = 3,83; F=0.054

4. Secondary Outcome: Staggered Spondaic Word Test
Description: Dichotic listening test in which two spondaic words are presented, one to each ear of the listener, in an overlapping fashion such that the first syllable of the first word is presented in isolation, the second syllable of the first word is presented simultaneously with the first syllable of the second word, and the second syllable of the second word is presented in isolation. Total number of test spondee pairs = 40.
Time Frame: Immediately post-intervention between weeks 8 and 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total errors
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
total errors | 5.1 (5.5) | 2.6 (2.7) | 5.2 (8.6) | 5.3 (6.6)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.554, ANOVA — df = 3,83; F=0.701

5. Secondary Outcome: Digit Span Score Measure of Auditory Working Memory
Description: The Digit Span subtest of the Wechsler Adult Intelligence Scale 3rd edition (WAIS-III) assessed auditory working memory. It consists of a Digit Span Forward task in which individuals to repeat numbers in the same sequence as they were presented verbally, and a Digit Span Backward task in which individuals repeat back the numbers in the reverse order to which they were heard. Data are summed to compute a Digit Span total score. Possible range of scores is 0 to 30, with higher scores indicating better performance.
Time Frame: Immediately post-intervention between weeks 8 and 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
units on a scale | 16 (5.0) | 17.5 (3.5) | 16.1 (4.6) | 16.4 (3.3)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.757, ANOVA — df = 3,83; F=0.395

6. Secondary Outcome: Time Compressed Speech Test (TCST)
Description: the TCST assessed speech recognition for speeded speech. Sentences are presented in the sound field in quiet at with 50% and 60% time compression. Participants repeat back each sentence after it is presented.
Time Frame: Immediately post-intervention between weeks 8 and 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
percent correct | 92.8 (4.6) | 93.8 (3.8) | 89.5 (9.7) | 90.9 (9.3)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.302, ANOVA; df = 3,83; F=1.236

7. Secondary Outcome: Cognitive Self Report Questionnaire (CSRQ).
Description: CSRQ assesses self-reported cognitive difficulties in 8 domains: Attention, Executive function, Memory, Language, Vision, Hearing, Energy,and Satisfaction. Participants respond on a 3-point Likert scale whether they perceived they improved, remained the same, or got worse as a result of an intervention. Total score is computed by summing scores on each subscale. Range for total score = -64 to +64, with higher scores indicating fewer reported cognitive difficulties.
Time Frame: Immediately post-intervention between weeks 8 and 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
units on a scale | 11.5 (14.1) | 10.3 (12.0) | 17.1 (16.1) | 0 (18.9)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.001, ANOVA; df = 3,83. F=6.343
Statistical Analysis 2: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: Speech, Spatial and Qualities of Hearing Scale-comparative (SSQ-C)
Description: Three subscale questionnaire that examines reported change in auditory disability for Speech, Spatial hearing and Quality of sounds. Subjects respond on a scale of -5 ('much worse') to +5 (much better) to indicate the change in difficulties following an intervention they have hearing in specific situations, with a lower number indicating greater difficulty. Results are presented for average total SSQ-C score which can range from -5 to +5, with higher scores indicating greater improvement.
Time Frame: Immediately post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Number analyzed (Participants) | 24 | 14 | 20 | 22
units on a scale | 1.0 (1.2) | 0.4 (0.6) | 1.0 (1.1) | 0.3 (0.7)
Statistical Analysis 1: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.013, ANOVA; df = 3,83; F=3.797
Statistical Analysis 2: Comparison: FM System vs Auditory Training vs FM System + Auditory Training vs Standard-of-care; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | FM System | Auditory Training | FM System + Auditory Training | Standard-of-care
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FM System (N=25) | Auditory Training (N=25) | FM System + Auditory Training (N=24) | Standard-of-care (N=25)
Participant reported mild headache following research visit at week 8 (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant reported headache after test session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes